CLINICAL TRIAL: NCT06610812
Title: KETOGENIC MEDITERRANEAN VERSUS HYPOCALORIC BALANCED DIET ON Added to Aerobic Exercises POLYCYSTIC OVARIAN ADOLESCENTS
Brief Title: "KETOGENIC MEDITERRANEAN VERSUS HYPOCALORIC BALANCED DIET ON POLYCYSTIC OVARIAN ADOLESCENTS"
Acronym: keto- MEDITERR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, shaimaa Mohamed hamed, Lecturer of physical therapy for women's health in MTIU, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo university
Record Dates: First submitted 2024-09-21; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Polycystic Ovary Disease
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled trail
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KETOGENIC MEDITERRANEAN diet (Experimental): It was consist of 20 adolescent females suffering from polycystic ovary disease. they received ketogenic Mediterranean diet program for 3 months with moderate aerobic exercises in the form of walking from 30 to 45 minutes a day, 3 times per week for 3 months.
  Interventions: Behavioral: KETOGENIC MEDITERRANEAN diet; Behavioral: moderate aerobic exercises
- HYPOCALORIC BALANCED DIET (Experimental): It was consist of 20 adolescent females suffering from polycystic ovary disease. they received hypo-caloric balanced diet program for 3 months with moderate aerobic exercises in the form of walking from 30 to 45 minutes a day, 3 times per week for 3 months.
  Interventions: Behavioral: hypo-caloric diet:; Behavioral: moderate aerobic exercises

INTERVENTIONS:
Behavioral: KETOGENIC MEDITERRANEAN diet — each patient in group A was instructed briefly about the nature of the treatment regimen to gain the patient's confidence and cooperation. the patient will receive ketogenic Mediterranean diet with aerobic training program. The diet will contain approximately 9300 kJ accordingly, 37% as total fat, 18% as monounsaturated and 9% as saturated, and 33 g of fiber per day for 3 months with moderate aerobic exercises in the form of walking from 30 to 45 minutes a day, 3 times per week for 3 months.
  This procedure performed by using the components of ketogenic Mediterranean diet:
  * Protein source: fatty fish, seafood, poultry, and eggs.
  * Fats and oils: olive oil, avocado oil, and MCT oil (medium-chain triglycerides oil).
  * Low carb vegetables: leafy greens, cruciferous vegetables, and other low carb veggies.
  * Low carb fruits: avocados, olives, and tomato.
  * Flavourings: paprika, cumin, cinnamon, coriander, anise, lemon or lime juice , mint , parsley and garlic .
  Other Names: KETO- MEDITERRANEAN
  Arms: KETOGENIC MEDITERRANEAN diet
Behavioral: hypo-caloric diet: — Group (b) received low caloric balanced diet regimen with aerobic exercise for 3 months in the form of moderate aerobic exercises in the form of walking for 30 to 45 minutes a day, 3 times per week for 3 months. This group received a diet of 1800 calories or lower accordingly including a combination of two or more of the following in each meal: Non starchy vegetable: spinach, broccoli, cauliflower, peppers, mushrooms, tomatoes, etc.
  Fruits: berries, apples bears, citrus fruits, melon, grapes bananas, etc. Starchy vegetables: potatoes peas, sweet potatoes etc. Fish and shellfish: salmon, clams, Trouts, oysters, etc. Eggs: whole eggs are more nutrient dense than white eggs. Poultry and meat: chicken turkey, beef, lamb, etc. Whole grains: oats, brown rice, farro etc. Legumes: chickpeas, kidney beans, lentils etc. Healthy fats: avocados, olive oil, unsweetened coconut, avocado oil. Dairy products: full-fat or reduced fat plain yogurt kefir and full-fat cheese.
  Other Names: hypo-caloric balanced diet:
  Arms: HYPOCALORIC BALANCED DIET
Behavioral: moderate aerobic exercises — moderate aerobic exercises in the form of walking from 30 to 45 minutes a day, 3 times per week for 3 months.
  Other Names: aerobic exercises

SUMMARY:
study was designed to determine the effect of ketogenic Mediterranean diet versus hypocaloric balanced diet on adolescent female with polycystic ovary disease.

DETAILED DESCRIPTION:
this study wsa designed to investigate the effect of the ketogenic Mediterranean diet in comparison with hypo-caloric diet on obese adolescent female's patients with polycystic ovary disease trying to find out a new physical therapy approach that had positive effect in the treatment and care for such cases which could enhance the physical therapy field.

ELIGIBILITY:
Inclusion Criteria:

1 - All patients were adolescent females. 2- All patients ages ranged from 16 to 21years old. 3- Their BMI ranged from 25kg/m² to 35kg/m². 4- All patients were suffering from hormonal disturbances confirmed by their lab tests and cysts in the ovaries that confirm their diagnosis with polycystic ovary disease.

5- They were conscious and free from any other medical disease.

Exclusion Criteria:

Patients were examined by a gynecologist before the study and excluded if they have:

1. Cardiac problems, epileptics and implanted pacemakers.
2. Pregnancy.
3. Malignancy and cardiovascular disease.
4. Women with skin infection.
5. Dysesthesia.
6. Cerebrovascular disease.
7. Uncontrolled diabetes.
8. Severe uncontrolled cardiac patient.
9. Liver and kidney dysfunction.

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — polycystic ovary disease
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-13 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
LH/FSH | 3 months
  Blood sample was taken from each woman before starting the study to measure the level of androgen in the blood and LH/FSH which will be estimated again after 3months to its level after each type of diet
body mass index | 3 months
  Weight and height measured while the patient is wearing a thin layer of clothes to calculate the body mass index according to the following equation in both groups: BMI=weight/height2 (Kg/m2)

SECONDARY OUTCOMES:
waist-hip ratio | 3 months
  A tape measurement wase used to determine the hip and waist circumference of each patient to calculate the waist-hip ratio by dividing the waist reading over the hip reading (the waist circumference should be measured at the midpoint between the lower margin of the last palpable ribs and the top of the iliac crest , hip circumference obtained by measuring at the top of the iliac crest in case the waist is convex rather than concave, such as with different body types, and obesity, the waist may be measured at a horizontal level (2.5 cm) above the umbilicus .for both measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Unversity, Giza, Egypt